CLINICAL TRIAL: NCT03340597
Title: A Phase I, Open Label Study in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Varying Oral Dosing Regimens for F901318
Brief Title: Assessment of Varying Oral Dosing Regimens for F901318 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: F901318-01-13-17
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1; F901318 (10 days) (Experimental): F901318 : 10 days dosing orally
  Interventions: Drug: F901318
- A2; F901318 (Experimental): F901318 : 10 days dosing orally, alternative dosing regimen
  Interventions: Drug: F901318
- A3; F901318 (Experimental): F901318 : 10 days dosing orally, alternative dosing regimen
  Interventions: Drug: F901318
- A4; F901318 (Experimental): F901318 : 10 days dosing orally, alternative dosing regimen
  Interventions: Drug: F901318

INTERVENTIONS:
Drug: F901318 — F901318 tablet

SUMMARY:
A Phase I, open label study evaluating safety, tolerability and pharmacokinetics of F901318 in healthy subjects following up to 28 days dosing, where F901318 is given orally . The effect of food upon the pharmacokinetics of F901318 and the effect of F901318 upon the pharmacokinetics of midazolam will also be assessed.

DETAILED DESCRIPTION:
Each cohort will comprise 12 healthy subjects and cohorts A1 (A2), B1 and B2 will be conducted in a sequential manner such that the dose level can be optimised upon review of emerging safety, tolerability and PK data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males or females of any ethnic origin between 18 and 55 years of age, weighing between 60 and 100 kg, with a body mass index (BMI) between 18 and 30 kg/m2.
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinaemia is not acceptable)
* Male subjects and female subjects of childbearing potential must agree to use appropriate contraception from screening, during the study and for 3 months after the last dose of study drug

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Subjects who have received any prescribed systemic or topical medication (other than hormonal contraception or hormone replacement therapy) within 14 days of the dose administration unless in the opinion of the Investigator and the medical monitor the medication will not interfere with the study procedures or compromise safety.
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator and the medical monitor the medication will not interfere with the study procedures or compromise safety.
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration unless in the opinion of the Investigator and the medical monitor the medication will not interfere with the study procedures or compromise safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 18 days
  safety and tolerability

SECONDARY OUTCOMES:
Area under the curve (AUC) 0-tau for F901318 | 11 days
  Pharmacokinetics (PK) of oral doses of F90318
maximum plasma concentration (Cmax) for F901318 | 11 days
  PK of oral doses of F90318
minimum plasma concentration (Cmin) for F901318 | 11 days
  PK of oral doses of F90318

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MB ChB PhD MRCS FFPM, Principal Investigator — Covance CRU Ltd
Locations (1):
- Covance Clinical Research Unit, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No